CLINICAL TRIAL: NCT05633550
Title: Evaluating the Test-retest Reliability of a Standardized Flexion - Extension Radiograph Imaging Protocol for the Lumbar Spine.
Brief Title: Flexion-Extension Radiograph Imaging Protocol Reliability Study
Status: Active, not recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: NL82684.091.22
Record Dates: First submitted 2022-11-10; First posted 2022-12-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Spinal Stenosis; Spinal Instability
Keywords: Diagnostic Imaging; Decision Support Systems, Clinical; Radiographic Image Interpretation, Computer-Assisted; Surgical Decompression
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flexion-extension radiographs — Participants will undergo (regular) flexion-extension radiographs.

SUMMARY:
Orthopedic surgeons often face the dilemma of whether to add fusion to a decompression procedure of the spine. Their decision mainly relies on personal experience to determine if a level is unstable preoperatively or if a specific decompression procedure might destabilize the spine. Lumbar spine flexion-extension radiographs aim to provide clinicians with images to assess the dynamism of a vertebral level, which crucial for evaluating spinal instability. However, the lack of a standardized imaging protocol for taking such flexion-extension radiographs leads to wide variability in their quality. This impacts the efficacy of radiographic measurements of angular and translational motion used for diagnosis. To effectively and reliably diagnose instability, it is crucial to control and standardize the flexion-extension radiograph protocols to promote the repeatability of intervertebral motion that characterizes a patient's full range of motion. The objective of this study is to evaluate the test-retest reliability of a standardized flexion - extension radiograph imaging protocol for the lumbar spine. This is an exploratory reliability study. A non-probability purposive sample of 45 patients with back pain from two tertiary care hospitals in The Netherlands is used. There is bo intervention. The main study parameter/endpoint is the agreement between the participants' first ("test") and second ("retest") kinematic results from their lumbar flexion-extension radiographs.

DETAILED DESCRIPTION:
Lumbar spinal stenosis, a narrowing of the spinal canal in the lower part of the back, is a relatively common medical problem, but optimal treatment for the condition is poorly understood. Lumbar spinal stenosis is commonly treated with decompression surgery (providing more space for the compressed nerve roots) with or without additional lumbar fusion surgery (connecting two or more vertebrae to eliminate instability). Orthopaedic surgeons are currently faced with the dilemma of whether or not to add fusion to a decompression procedure. To decide between these two surgical options, surgeons rely mostly on their personal experience. They have to subjectively gauge whether a level is unstable preoperatively or if a specific decompression procedure is likely to destabilize the spine. A valid and reliable test for spinal instability would facilitate research to determine whether spinal instability measurements can be used to choose the optimal surgical treatment for each level.

A reliable diagnostic assessment for spinal instability would ideally be validated using an existing "gold standard" test. Such a test should have a very high sensitivity and specificity and must be supported by clearly developed rationale and high-quality evidence. Unfortunately, such a test does not currently exist for spinal instability. However, abnormalities in intervertebral motion are often a hallmark for spinal instability. A commonly accepted way to examine intervertebral motion is by analyzing the patient's flexion-extension radiographs. Using these two radiographs, the spine's sagittal plane intervertebral motion can be measured. The relative motion between the two images can be measured at all relevant levels either through manual measurement or computer assisted methods. Ideally, a standardized flexion-extension radiograph imaging protocol accomplishes the following: the patient sufficiently stresses the spine in order to assess the integrity of intervertebral motion restraints (ligaments, annulus, facet capsule, etc.), it is easily implemented into the clinical work flow, and it is reliable and repeatable across subjects and clinicians.

A myriad of patient positioning protocols for the flexion-extension radiograph imaging procedure have been tested and deployed, although generally without well-validated success criteria. Despite the large amount of studies on the topic, no one flexion-extension radiograph imaging protocol has been widely accepted. This suggests that 1) the studies were not appropriately powered to influence change, 2) some protocols (methods, equipment, instructions, etc.) are not easily implemented or practical in routine clinical workflows, 3) acquiring radiograph images of the lumbar spine in sufficiently stressed positions is not widely accepted as clinically important, or 4) most ordering clinicians do not realize how often a patient fails to adequately stress the spine while undergoing a standard of care flexion-extension radiograph. One factor that can often cast doubt on the efficacy of the flexion-extension radiograph procedure is the level of patient effort or range of spinal motion achieved by the patient. For standing flexion-extension radiographs, more patient effort leads to more intervertebral motion. This is a fairly simple and intuitive concept. However, achieving maximum patient effort is not a simple task. It could be argued that symptomatic patients should not be expected to exert maximum effort because it can be painful or uncomfortable. This argument can be supplemented with evidence that fear avoidance can limit motion and intervertertebral motion is substantially increased after analgesic injections.

Despite some of the arguments that can be used against the implementation of standardized flexion-extension radiograph imaging protocols in assessing spinal instability, there is ample data that good patient effort can be obtained in symptomatic patients. In one large multi-site study of lumbar stenosis with the exact same patient inclusion/exclusion criteria, a large amount of variance can be seen in the average level of intervertebral rotation. This suggests that differences in the flexion-extension radiograph protocol could be the driving factor in this high amount of variance seen between sites. It is also possible that the physician and/or radiology technician helped to quell patient's fear of motion by explaining that the maximum flexion and extension will not injure their back and will provide the best data for a reliable diagnosis.

With this in mind, the need for a standardized flexion-extension radiograph imaging protocol to assess for spinal instability is evident. Such standardized protocols can influence the amount of intervertebral motion, both translational and rotational. Since intervertebral motion is often used as evidence for spinal instability, inadequate effort likely leads to false negatives for spinal instability. Thus, developing a standardized imaging protocol to reliably measure intervertebral motion during a flexion-extension exam is clinically significant, as it often influences the diagnosis of a patient.

ELIGIBILITY:
Inclusion Criteria:

* referral to the orthopaedic surgeon because of pain in the back or leg and requiring lumbar spine radiographs so the orthopaedic surgeon is able to diagnose the probable cause of the pain.
* over the age of 18 years
* ability to flex and extend the spine sufficiently to facilitate acceptable flexion and extension radiographs.

Exclusion Criteria:

* any form of spine-related traumatic injury
* prior lumbar spinal surgery
* lateral spondylolisthesis or coronal plane curvature in the lumbar spine of >10°
* the presence of involuntary back muscle spasms
* the presence of significant changes in pain during the day
* inability to understand and sign the study Informed Consent form
* inability to follow oral instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A non-probability purposive sample of 45 patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between the participants' first ("test") and second ("retest") kinematic results: intervertebral translation, intervertebral rotation and a value derived form the latter: translation-per-degree-of-rotation. | One hour after taking both sets of the flexion-extension radiographs
  Test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Job LC van Susante, Dr. PhD., Principal Investigator — Department of orthopedics, Rijnstate Hospital
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - OLVG, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hipp JA, Guyer RD, Zigler JE, Ohnmeiss DD, Wharton ND. Development of a novel radiographic measure of lumbar instability and validation using the facet fluid sign. Int J Spine Surg. 2015 Jul 17;9:37. doi: 10.14444/2037. eCollection 2015. PMID 26273555
- [Background] Zhao K, Yang C, Zhao C, An KN. Assessment of non-invasive intervertebral motion measurements in the lumbar spine. J Biomech. 2005 Sep;38(9):1943-6. doi: 10.1016/j.jbiomech.2004.07.029. PMID 16023484
- [Background] Pearson AM, Spratt KF, Genuario J, McGough W, Kosman K, Lurie J, Sengupta DK. Precision of lumbar intervertebral measurements: does a computer-assisted technique improve reliability? Spine (Phila Pa 1976). 2011 Apr 1;36(7):572-80. doi: 10.1097/BRS.0b013e3181e11c13. PMID 21217439
- [Background] Patwardhan AG, Havey RM, Wharton ND, Tsitsopoulos PP, Newman P, Carandang G, Voronov LI. Asymmetric motion distribution between components of a mobile-core lumbar disc prosthesis: an explanation of unequal wear distribution in explanted CHARITE polyethylene cores. J Bone Joint Surg Am. 2012 May 2;94(9):846-54. doi: 10.2106/JBJS.J.00638. PMID 22552675
- [Background] Auerbach JD, Namdari S, Milby AH, White AP, Reddy SC, Lonner BS, Balderston RA. The parallax effect in the evaluation of range of motion in lumbar total disc replacement. SAS J. 2008 Dec 1;2(4):184-8. doi: 10.1016/SASJ-2008-0020-RR. eCollection 2008. PMID 25802620
- [Background] Zhao KD, Ben-Abraham EI, Magnuson DJ, Camp JJ, Berglund LJ, An KN, Bronfort G, Gay RE. Effect of Off-Axis Fluoroscopy Imaging on Two-Dimensional Kinematics in the Lumbar Spine: A Dynamic In Vitro Validation Study. J Biomech Eng. 2016 May;138(5):054502. doi: 10.1115/1.4032995. PMID 26974192
- [Background] Weiler PJ, King GJ, Gertzbein SD. Analysis of sagittal plane instability of the lumbar spine in vivo. Spine (Phila Pa 1976). 1990 Dec;15(12):1300-6. doi: 10.1097/00007632-199012000-00012. PMID 2149207
- [Background] Staub BN, Holman PJ, Reitman CA, Hipp J. Sagittal plane lumbar intervertebral motion during seated flexion-extension radiographs of 658 asymptomatic nondegenerated levels. J Neurosurg Spine. 2015 Dec;23(6):731-8. doi: 10.3171/2015.3.SPINE14898. Epub 2015 Aug 21. PMID 26296193
- [Background] Hasegawa K, Shimoda H, Kitahara K, Sasaki K, Homma T. What are the reliable radiological indicators of lumbar segmental instability? J Bone Joint Surg Br. 2011 May;93(5):650-7. doi: 10.1302/0301-620X.93B5.25520. PMID 21511932
- [Background] Bogduk, N., Instability, in Clinical and Radiological Anatomy of the Lumbar Spine, N. Bogduk, Editor. 2012, Elsevier Health Sciences. p. 207-216
- [Background] Hipp JA, Chan EF. Threshold Limit Graphical Approach to Understanding Outcome Predictive Metrics: Data from the Osteoarthritis Initiative. Cureus. 2017 Jul 8;9(7):e1447. doi: 10.7759/cureus.1447. PMID 29034136
- [Background] Cardis E, Vrijheid M, Blettner M, Gilbert E, Hakama M, Hill C, Howe G, Kaldor J, Muirhead CR, Schubauer-Berigan M, Yoshimura T, Bermann F, Cowper G, Fix J, Hacker C, Heinmiller B, Marshall M, Thierry-Chef I, Utterback D, Ahn YO, Amoros E, Ashmore P, Auvinen A, Bae JM, Solano JB, Biau A, Combalot E, Deboodt P, Diez Sacristan A, Eklof M, Engels H, Engholm G, Gulis G, Habib R, Holan K, Hyvonen H, Kerekes A, Kurtinaitis J, Malker H, Martuzzi M, Mastauskas A, Monnet A, Moser M, Pearce MS, Richardson DB, Rodriguez-Artalejo F, Rogel A, Tardy H, Telle-Lamberton M, Turai I, Usel M, Veress K. Risk of cancer after low doses of ionising radiation: retrospective cohort study in 15 countries. BMJ. 2005 Jul 9;331(7508):77. doi: 10.1136/bmj.38499.599861.E0. Epub 2005 Jun 29. PMID 15987704
- [Background] Bolus NE. NCRP report 160 and what it means for medical imaging and nuclear medicine. J Nucl Med Technol. 2013 Dec;41(4):255-60. doi: 10.2967/jnmt.113.128728. Epub 2013 Oct 31. PMID 24179182
- [Background] Transport, E.C.D.-G.f.E.a., European guidance on estimating population doses from medical x-ray procedures. 2008.
- [Background] Environment, E.C.D.-G.f., Guidance on medical exposures in medical and biomedical research. 1999, European Commission Publications Office.
- [Background] (NFU), N.F.v.U.M.C., Richtlijn Kwaliteitsborging Mensgebonden Onderzoek. 2020, Nederlandse Federatie van Universitair Medische Centra (NFU)
- [Background] JA, H., et al., A new method correlating an objective radiographic metric for lumbar spine instability and the facet fluid sign on MRI, in International Society of the Advancement of Spine Surgery. 2015: San Diego.
- [Background] Hipp, J., P. Newman, and O. Avila-Montes. Toward standardization of lumbar flexion-extension studies. in ISASS. 2018. Toronto